CLINICAL TRIAL: NCT05361265
Title: THE EFFECT OF FETAL MOVEMENT COUNTING ON PRENATAL MATERNAL ATTACHMENT AND DISTRESS IN PREGNANCY
Brief Title: FETAL MOVEMENT COUNTING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Şengül Yaman Sözbir, Assoc Prof, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HulyaAydin
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: the Effect of Fetal Movement Count on Prenatal Attachment and Pregnancy Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): pregnant women were trained about fetal movements and fetal movement counting was taught. The training was given verbally. Pregnant women were asked to perform ten fetal movements by counting once a day after any meal, lying in the left side position for one hour. When ten fetal movements could not be reached within the first hour, pregnant women were instructed to count the fetal movements for one hour after walking for five minutes. When ten fetal movement counts could not be obtained at the end of two hours, they were asked to apply to the hospital immediately. Pregnant women were expected to perform fetal movement counting after the same meal every day (breakfast, lunch or dinner) and record the start and end times of the ten movements on the Fetal Movement Monitoring Card.
  Interventions: Other: fetal movement counting
- Control Group (No Intervention): Routine follow up

INTERVENTIONS:
Other: fetal movement counting — pregnant women were trained about fetal movements and fetal movement counting was taught. Pregnant women were asked to perform ten fetal movements by counting once a day. In the application of the study, it was ensured that the pregnant women in the experimental group performed fetal movement counting for at least four to six weeks. In this context, pregnant women were called every week to monitor and to motivate them to continue the counting.
  Arms: Experimental Group

SUMMARY:
Purpose: This study aimed to determine the effect of fetal movement counting on prenatal maternal attachment and distress in pregnancy.

Methods: This is a quasi-experimental study. The population of the study consisted of of 60 primigravida pregnant women (30 experimental and 30 control groups) being in 28 to 32 weeks gestation. The Prenatal Attachment Inventory (PAI) and the Tilburg Pregnancy Distress Scale (TPDS) used for data collection. After the pre-tests (28 to 32 weeks gestation), the experimental group were trained about fetal movement counting. The experimental group performed fetal movement counting for at least four to six weeks. The post-tests were filled in 32 to 38 weeks gestation. The control group received only pre-tests and post-test in the same weeks gestation with the experimental group.

DETAILED DESCRIPTION:
This is a quasi-experimental study.

The population of the study consisted of pregnant women followed in a State Hospital in the capital city of Turkey in 2019. Power analysis (Sample error: 0.01 and power: 95%) was performed to determine the sample size of the study. In the power analysis, the mean score of the Prenatal Attachment Inventory was 71.88 ± 8.25 [15] and the mean score of the Tilburg Pregnancy Distress Scale was 18.86 ± 7.37 [16]. The minimum number of participants required for each group was 24 (α = 0.05, 1-β = 0.80). To increase the reliability and validity of the study, the study sample consisted of 60 pregnant women (30 experimental and 30 control groups). The criteria for inclusion in the research sample were; being in 28 to 32 weeks gestation, primigravity, being at least literate, not having any chronic or psychiatric disease, not having any communication disability (speech, hearing, mental), non-risky pregnancy (preeclampsia, gestational diabetes, advanced age, and adolescent pregnancy, etc.), current or recent pregnancy is identified as not having any significant life difficulties (loss, illness, accident, etc.). The experimental and control groups were matched to be similar in terms of age, education and working status parameters.

Data Collection Instruments:

Research data were collected using the Descriptive Information Form, the Prenatal Attachment Inventory (PAI), the Tilburg Pregnancy Distress Scale (TPDS) and the Fetal Movement Monitoring Card.

In the Descriptive Information Form, there are five questions including the socio-demographic informations of the pregnant women (age, education status, working status, and perceived income) and the gestational week.

The PAI was developed by Mary Muller (1993) to explain the feelings, thoughts, and situations of women during pregnancy and to determine their attachment levels to the baby in the prenatal period [17]. The scale consists of 21 items in total. In the 4-point Likert scale, each item can score between 1 and 4 points (1: Never, 2: Sometimes, 3: Frequent, 4: Always). The highest score of the scale is 84, the lowest score is 21, and the high scale score indicates the high level of prenatal attachment. The Turkish reliability and validity study of the scale was conducted by Duyan et al. (2013) and the Cronbach Alpha reliability coefficient was found to be 0.78 [18]. In our study, Cronbach Alpha reliability coefficients were; pre-test: 0.851, post-test: 0.811 in the experimental group; pre-test: 0.863, post-test: 0.865 in control group.

The TPDS is developed by Pop et al. (2011) for the diagnosis of distress in pregnancy [11]. The scale consists of a total of 16 items. The scale has two subscales. Negative Affect subscale consists of 12 items including fear, anxiety and negative perceptions regarding pregnancy, childbirth and the postpartum period. Partner Involvement subscale consists of 4 items related to spousal support during pregnancy. The scale is a four-point Likert type and each item is scored between 1 and 3 (0: very often, 1: quite often, 2: sometimes, and 3: rarely or never). The points 3.5,6,7,9,10,11,12,13,14 and 16 are interpreted by reversing them. The highest score of the scale is 48 and the lowest score is 0. A high score from the scale indicates that pregnant women are at risk for distress. The Turkish validity-reliability study of the scale was conducted by Çapık and Pasinlioğlu (2015) and the Cronbach Alpha reliability coefficient was found to be 0.83 [19]. In our study, the Cronbach's alpha reliability coefficient of the scale was 0.836 in the experimental group and 0.826 in the post-test; the control group's pre-test was 0.731 and the post-test was 0.793.

The Fetal Movement Monitoring Card was prepared by the researchers. The card contains instructions on the importance of fetal movement counting and information on how to perform the counting. The card also includes a chart to monitor the fetal movement counting process performed by pregnant women and record the fetal movement counting process and how many movements are counted to check whether the researcher fulfilled the research conditions of the pregnant women.

Procedure:

Ethics committee approval and hospital permissions were obtained for the study. The application was carried out in the pregnant education class of the hospital between 01.11.2018-18.02.2019. It was determined that the pregnant women who participated in the pregnant education class met the research criteria. Written consent was obtained after the pregnant women who met the criteria were informed about the study. The pregnant women were assigned to the experimental and control groups by the researcher. At this stage of the study, all data collection forms were filled out for pregnant women. The forms were completed by the pregnant women themselves in a comfortable environment in a quiet part of the pregnant education class.

Control Group:

When the pregnant women in the control group came to the hospital for follow-up (in 32 to 38 weeks gestation), they were invited to the pregnant education class and the PAI and the TPDS was refilled.

Experimental Group:

After completing the data collection tools, pregnant women were trained about fetal movements and fetal movement counting was taught. The training was given verbally. Pregnant women were asked to perform ten fetal movements by counting once a day after any meal, lying in the left side position for one hour. When ten fetal movements could not be reached within the first hour, pregnant women were instructed to count the fetal movements for one hour after walking for five minutes. When ten fetal movement counts could not be obtained at the end of two hours, they were asked to apply to the hospital immediately. Pregnant women were expected to perform fetal movement counting after the same meal every day (breakfast, lunch or dinner) and record the start and end times of the ten movements on the Fetal Movement Monitoring Card.

In the application of the study, it was ensured that the pregnant women in the experimental group performed fetal movement counting for at least four to six weeks. In this context, pregnant women were called every week to monitor and to motivate them to continue the counting. It was planned to exclude the pregnant women who were informed that they had not performed the application for four consecutive days, withdrew from the study voluntarily, who could not be followed up by telephone, who had significant life distress (death, illness, divorce, accident, etc.), who developed complications in their pregnancy or was diagnosed with risky pregnancy. In this context, one pregnant was excluded from the sample because she gave birth prematurely and two pregnant women did not answer the phone. New pregnant women who met the criteria were included in the sample instead of the pregnant women outside the sample.

When the pregnant women came to the hospital for follow-up (in 32 to 38 weeks gestation), they were invited to the pregnant education class. After confirming that the women had performed the application by checking the Fetal Movement Monitoring Cards, the API and the TPDS were refilled.

ELIGIBILITY:
Inclusion Criteria:

* being in 28 to 32 gestation weeks
* primigravidity
* at least literate

Exclusion Criteria:

* illiteration
* chronic or psychiatric disease
* communication disability (speech, hearing, mental)
* risky pregnancy

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
prenatal maternal attachment | 4-6 weeks
  the Prenatal Attachment Inventory: The inventory was developed to explain the feelings, thoughts, and situations of women during pregnancy and to determine their attachment levels to the baby in the prenatal period [17]. The scale consists of 21 items in total. In the 4-point Likert scale, each item can score between 1 and 4 points (1: Never, 2: Sometimes, 3: Frequent, 4: Always). The highest score of the scale is 84, the lowest score is 21, and the high scale score indicates the high level of prenatal attachment.
distress in pregnancy | 4-6 weeks
  the Tilburg Pregnancy Distress Scale: The scale was developed for the diagnosis of distress in pregnancy [11]. The scale consists of a total of 16 items. The scale has two subscales. Negative Affect subscale consists of 12 items including fear, anxiety and negative perceptions regarding pregnancy, childbirth and the postpartum period. Partner Involvement subscale consists of 4 items related to spousal support during pregnancy. The scale is a four-point Likert type and each item is scored between 1 and 3 (0: very often, 1: quite often, 2: sometimes, and 3: rarely or never). The points 3.5,6,7,9,10,11,12,13,14 and 16 are interpreted by reversing them. The highest score of the scale is 48 and the lowest score is 0. A high score from the scale indicates that pregnant women are at risk for distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No